CLINICAL TRIAL: NCT03966157
Title: The Role of a Nasal Bridle in the Frequency of Repeat Endoscopic Procedures for Endoscopic Naso-enteric Tube Placement
Brief Title: Nasal Bridles and Repeat Endoscopic Procedures for Endoscopic Nasoenteric Tubes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: St. Louis University (Other)
Responsible Party: Principal Investigator, Samuel Burton, MD, Gastroenterology Fellow, St. Louis University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 29703
Record Dates: First submitted 2019-05-22; First posted 2019-05-29 (Actual); Results first posted 2023-05-19 (Actual); Last update posted 2023-05-19 (Actual); Status verified 2023-05

CONDITIONS: Feeding Disorders
MeSH Terms: conditions — Feeding and Eating Disorders

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Nasal Bridle (Experimental): Patients randomized to have nasal bridle.
  Interventions: Device: Nasal Bridle
- Standard (No Intervention): Patients randomized with adhesive tape.

INTERVENTIONS:
Device: Nasal Bridle — Feeding tube secured with nasal bridle
  Arms: Nasal Bridle

SUMMARY:
In critically ill patients, nutrition is a major part of healing and recovery. In patients unable to tolerate oral feeding, nasoenteric tube feeding (a tube placed from the nose to the stomach or small intestine) provides a safe alternative for feeding. Some patients require these tubes to be placed endoscopically due to numerous patient factors including difficult anatomy, need for post-gastric feeding, among others). In patients that require endoscopically placed tubes, there is risk of perforation, infection, bleeding, aspiration, and rarely even death. In patients that have recurrent dislodgement of endoscopically placed tubes, the need for repeat endoscopy increases patient exposure to these risks. Traditional securing mechanism with adhesive tape to reduce dislodgment often fail in critically ill patients requiring patients to have repeat endoscopies to replace nasoenteric feeding tubes and subjects patients potentially to increased cumulative risks associated with each endoscopy.

The investigators propose to collect data for one year, the investigators will prospectively follow via chart review endoscopically placed naso-enteric tubes placed with a Standard AMT Bridle securement device and assess if there is a reduction in accidental tube removal requiring replacement endoscopically.

DETAILED DESCRIPTION:
Patients to be recruited are those who are scheduled to undergo routine upper endoscopy with nasoenteric tube placement. Patients will be randomized into two groups: control arm and device arm.

Control arm includes patients that will have nasoenteric tubes secured with standard protocol, adhesive tape. Device arm includes patients that will have nasoenteric tubes secured with Standard AMT Bridle. The nasal bridles will be placed by the endoscopist. Upper endoscopy will not be affected. Placement of nasal bridle will take 1-2 minutes after endoscopic procedure completed. No addition sedation, medication or exposure necessary.

Patients will be randomized by sealed envelope randomization. Clinicians are given randomly generated treatment allocations within sealed opaque envelopes. Once a patient has consented to enter the study trial an envelope is opened and the patient is then offered the allocated treatment regimen. Patients will be consented by a member of the research team prior to endoscopy. Randomization will be singly blinded only to the the patient prior to endoscopy. Endoscopist will not be blinded as they will be placing the securement device and in order to reduce selection bias.

In the event of tube dislodgment, the patient will receive same treatment.

Follow-up of patients will occur via chart review until the time of discharge, at 6 months and at 12 months after feeding tube placement via chart review. Data collected with include repeat EGD, length of endoscopy, length of hospital stay, and mortality. The number of endoscopies and repeated nasoenteric tubes placed will be tracked at six and twelve months.

ELIGIBILITY:
Inclusion Criteria:

* Patients in need for endoscopically placed nasoenteric feeding tube

Exclusion Criteria:

* Age greater than 90 years

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2019-06-19 (Actual); Primary Completion 2022-03-25 (Actual); Study Completion 2022-03-25 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Samuel Burton, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Nasal Bridle | Standard
Started | 17 | 14
Completed | 16 | 14
Not Completed | 1 | 0
Not completed — Physician Decision | 1 | 0

BASELINE CHARACTERISTICS:
Population: One patient randomized to nasal bridle, but did not complete study as there was change in clinical status
Groups:
- Total: Total of all reporting groups
Arm/Group | Nasal Bridle | Standard | Total
Number analyzed (Participants) | 16 | 14 | 30
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 13 | 11 | 24
  >=65 years | 3 | 3 | 6
Age, Continuous [Mean (Full Range); unit: years] | 54.8 [18 to 77] | 53.4 [31 to 82] | 54.0 [18 to 82]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 7 | 16
  Male | 7 | 7 | 14
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 16 | 14 | 30

OUTCOME MEASURES:

1. Primary Outcome: Repeat Endoscopy to Replace Dislodged Feeding Tube
Description: The number of participants that require a repeat endoscopy to place an additional nasoenteric tube due to inadvertent dislodgement
Time Frame: 12 months
Population: One patient randomized to nasal bridle completed procedure but was lost to follow-up
Measure: Count of Participants; unit: Participants
Arm/Group | Nasal Bridle | Standard
Number analyzed (Participants) | 15 | 14
Participants | 3 | 2

2. Secondary Outcome: Inadvertent Tube Dislodgement
Description: Number of participants that inadvertently have nasoenteric tube dislodged
Time Frame: 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | Nasal Bridle | Standard
Number analyzed (Participants) | 15 | 14
Participants | 7 | 2

ADVERSE EVENTS:
Time Frame: 1 year
Groups:
- Nasal Bridle: Patients randomized to nasal bridle.
Arm/Group | Nasal Bridle | Standard
All-Cause Mortality (participants affected / at risk) | 0/16 | 0/14
Serious Adverse Events (participants affected / at risk) | 0/16 | 0/14
Other Adverse Events (participants affected / at risk) | 0/16 | 0/14

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-06-13): https://cdn.clinicaltrials.gov/large-docs/57/NCT03966157/Prot_SAP_001.pdf